CLINICAL TRIAL: NCT00491179
Title: Retreatment of Dialysis Patients With Chronic Hepatitis C With Pegylated Interferon Alfa-2a Plus Low Dose Ribavirin Who Fail Interferon Alfa or Pegylated Interferon Alfa Monotherapy - a Pilot Study
Brief Title: Retreatment of Dialysis Patients With Chronic Hepatitis C With Pegylated Interferon Alfa-2a Plus Low Dose Ribavirin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Dr. Chen-Hua Liu, National Taiwan University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200703032M
Record Dates: First submitted 2007-06-23; First posted 2007-06-26 (Estimated); Results first posted 2009-11-13 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-10

CONDITIONS: Chronic Hepatitis C; Hemodialysis
Keywords: Chronic hepatitis C; hemodialysis; interferon; ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pegylated IFN + RBV for HCV genotype 1 (Experimental): Pegylated interferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 135 ug/week plus ribavirin (Copegus, F. Hoffman-LaRoche) 200 mg/day for 48 weeks for HCV genotype 1
  Interventions: Drug: Pegylated interferon alfa-2a and ribavirin
- Pegylated IFN + RBV for HCV genotype 2 (Experimental): Pegylated interferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 135 ug/week plus ribavirin (Copegus, F. Hoffman-LaRoche) 200 mg/day for 24 weeks for HCV genotype 2
  Interventions: Drug: Pegylated interferon alfa-2a and ribavirin

INTERVENTIONS:
Drug: Pegylated interferon alfa-2a and ribavirin — Pegylated interferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 135 ug/week plus ribavirin (Copegus, F. Hoffman-LaRoche) 200 mg/day for 48 weeks
  Arms: Pegylated IFN + RBV for HCV genotype 1
Drug: Pegylated interferon alfa-2a and ribavirin — Pegylated interferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 135 ug/week plus ribavirin (Copegus, F. Hoffman-LaRoche) 200 mg/day for 24 weeks
  Arms: Pegylated IFN + RBV for HCV genotype 2

SUMMARY:
Chronic hepatitis C virus (HCV) infection is common in dialysis patients. Interferon (IFN)-based treatment for chronic hepatitis C has been the mainstay therapy in immunocompetent patients. Two meta-analyses evaluating the efficacy and safety of conventional IFN alfa monotherapy showed that the sustained virologic response (SVR) rates were 37% and 33%, respectively; and the corresponding dropout rates were 17% and 29.6%, respectively. The efficacy and safety of pegylated IFN alfa-2a and 2b in treating dialysis patients showed conflicting results, with a more favorable outcome of patients treated with pegylated IFN alfa-2a (135-180 μg/week: SVR 33-75%, well tolerated) than those treated with pegylated IFN alfa-2b (0.5-1.0 μg/week: SVR 12.5%, poorly tolerated), Currently, IFN-based therapy to treatment HCV infection should be initiated in dialysis stages, because the use of IFN in RT patients harbors high risks of acute graft rejection,and have low response rates under the concomitant use of immunosuppressive agents.

Ribavirin, which has been used in combination with IFN to treat chronic hepatitis C in the general patients and achieve a higher SVR rate than IFN monotherapy, is considered contraindicated in dialysis patients with chronic hepatitis C due to the risk of severe hemolytic anemia. However, some pilot studies evaluating combined conventional IFN alfa plus low dose ribavirin (170-300 mg/day) showed SVR rates of 17%-66% after 24-48 weeks of treatment.In addition, a recent study including 6 patients with combination of pegylated IFN alfa plus low dose ribavirin also showed a SVR rate of 50%.

Although dialysis patients have a higher SVR rate to conventional IFN or pegylated IFN monotherapy than patients with normal renal function for HCV therapy. More than half of these patients are relapsers or non-responders to IFN monotherapy. Retreatment of HCV-patients with normal renal function by combined pegylated IFN alfa plus ribavirin who fail to response to IFN monotherapy has achieved a SVR rate of 28%. Based on the long-term favorable outcome in dialysis patients who eradicate HCV, the aim of the study is to evaluate the efficacy and safety of retreatment by pegylated IFN alfa-2a plus low dose ribavirin in dialysis patients who fail to achieve HCV eradication by conventional or pegylated IFN alfa.

DETAILED DESCRIPTION:
Chronic hepatitis C virus (HCV) infection is common in dialysis patients, with the reported prevalence varying from 3% to 80% worldwide.(1-3) Although these patients usually have mild symptoms and moderate elevation of alanine transaminase levels, recent international collaborative survey and prospective studies found that anti-HCV seropositivity and positive HCV RNA were risk factors for mortality and hepatocellular carcinoma (HCC).(4-7) Furthermore, progressive hepatic fibrosis, poor patient and graft survival were observer in dialysis patients with HCV infection who undergo renal transplantation (RT), suggesting immunosuppression following RT may worsen the course of hepatic fibrosis and renal graft function.(8-13) These lines of evidence indicate that HCV infection in the dialysis population is an important issue to be tackled.

Interferon (IFN)-based treatment for chronic hepatitis C has been the mainstay therapy in immunocompetent patients. In dialysis patients, treatment with conventional or pegylated interferon has also received much attention recently. Two meta-analyses evaluating the efficacy and safety of conventional IFN alfa monotherapy showed that the sustained virologic response (SVR) rates were 37% and 33%, respectively; and the corresponding dropout rates were 17% and 29.6%, respectively.(14,15) The efficacy and safety of pegylated IFN alfa-2a and 2b in treating dialysis patients showed conflicting results, with a more favorable outcome of patients treated with pegylated IFN alfa-2a (135-180 μg/week: SVR 33-75%, well tolerated) than those treated with pegylated IFN alfa-2b (0.5-1.0 μg/week: SVR 12.5%, poorly tolerated),(16-21) which may result from different pharmacokinetic profiles between these two pegylated IFNs. Currently, IFN-based therapy to treatment HCV infection should be initiated in dialysis stages, because the use of IFN in RT patients harbors high risks of acute graft rejection,(22,23) and have low response rates under the concomitant use of immunosuppressive agents.(24,25) Ribavirin, which has been used in combination with IFN to treat chronic hepatitis C in the general patients and achieve a higher SVR rate than IFN monotherapy, is considered contraindicated in dialysis patients with chronic hepatitis C due to the risk of severe hemolytic anemia. However, some pilot studies evaluating combined conventional IFN alfa plus low dose ribavirin (170-300 mg/day) showed SVR rates of 17%-66% after 24-48 weeks of treatment.(26-28) In addition, a recent study including 6 patients with combination of pegylated IFN alfa plus low dose ribavirin also showed a SVR rate of 50%.(29) Although dialysis patients have a higher SVR rate to conventional IFN or pegylated IFN monotherapy than patients with normal renal function for HCV therapy. More than half of these patients are relapsers or non-responders to IFN monotherapy. Retreatment of HCV-patients with normal renal function by combined pegylated IFN alfa plus ribavirin who fail to response to IFN monotherapy has achieved a SVR rate of 28%.(30) Based on the long-term favorable outcome in dialysis patients who eradicate HCV, the aim of the study is to evaluate the efficacy and safety of retreatment by pegylated IFN alfa-2a plus low dose ribavirin in dialysis patients who fail to achieve HCV eradication by conventional or pegylated IFN alfa.

ELIGIBILITY:
Inclusion Criteria:

* Non-responders or relapsers of dialysis patients to conventional interferon or pegylated interferon monotherapy
* Age 18~65 years old
* Creatinine clearance (Ccr) < 10 ml/min/1.73 m2
* Anti-HCV (Abbott HCV EIA 2.0, Abbott Diagnostic, Chicago, IL) positive > 6 months
* Detectable serum quantitative HCV-RNA (Cobas Taqman HCV Monitor v2.0, Roche Diagnostics) with dynamic range 25- 391000000 IU/ml

Exclusion Criteria:

* Severe anemia (hemoglobin < 10 g/dL) or hemoglobinopathy
* Neutropenia (neutrophil count, <1,500/mm3)
* Thrombocytopenia (platelet <90,000/ mm3)
* Co-infection with HBV or HIV
* Chronic alcohol abuse (daily consumption > 20 g/day)
* Autoimmune liver disease
* Decompensated liver disease (Child classification B or C)
* Neoplastic disease
* An organ transplant
* Immunosuppressive therapy
* Poorly controlled autoimmune diseases, pulmonary diseases, cardiac diseases, psychiatric diseases, neurological diseases, diabetes mellitus
* Evidence of drug abuse
* Unwilling to have contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-06; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hua Liu, MD, Study Chair — Department of Internal Medicine, National Taiwan Universitys Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Fabrizi F, Poordad FF, Martin P. Hepatitis C infection and the patient with end-stage renal disease. Hepatology. 2002 Jul;36(1):3-10. doi: 10.1053/jhep.2002.34613. PMID 12085342
- [Background] Kao JH, Huang CH, Chen W, Tsai TJ, Lee SH, Hung KY, Chen DS. GB virus C infection in hemodialysis patients: molecular evidence for nosocomial transmission. J Infect Dis. 1999 Jul;180(1):191-4. doi: 10.1086/314850. PMID 10353878
- [Background] Hou CH, Chen WY, Kao JH, Chen DS, Yang Y, Chen JJ, Lee SH, Wu DJ, Yang SC. Intrafamilial transmission of hepatitis C virus in hemodialysis patients. J Med Virol. 1995 Apr;45(4):381-5. doi: 10.1002/jmv.1890450405. PMID 7545208
- [Background] Maisonneuve P, Agodoa L, Gellert R, Stewart JH, Buccianti G, Lowenfels AB, Wolfe RA, Jones E, Disney AP, Briggs D, McCredie M, Boyle P. Cancer in patients on dialysis for end-stage renal disease: an international collaborative study. Lancet. 1999 Jul 10;354(9173):93-9. doi: 10.1016/s0140-6736(99)06154-1. PMID 10408483
- [Background] Nakayama E, Akiba T, Marumo F, Sato C. Prognosis of anti-hepatitis C virus antibody-positive patients on regular hemodialysis therapy. J Am Soc Nephrol. 2000 Oct;11(10):1896-1902. doi: 10.1681/ASN.V11101896. PMID 11004221
- [Background] Stehman-Breen CO, Emerson S, Gretch D, Johnson RJ. Risk of death among chronic dialysis patients infected with hepatitis C virus. Am J Kidney Dis. 1998 Oct;32(4):629-34. doi: 10.1016/s0272-6386(98)70027-7. PMID 9774125
- [Background] Pereira BJ, Natov SN, Bouthot BA, Murthy BV, Ruthazer R, Schmid CH, Levey AS. Effects of hepatitis C infection and renal transplantation on survival in end-stage renal disease. The New England Organ Bank Hepatitis C Study Group. Kidney Int. 1998 May;53(5):1374-81. doi: 10.1046/j.1523-1755.1998.00883.x. PMID 9573555
- [Background] Mathurin P, Mouquet C, Poynard T, Sylla C, Benalia H, Fretz C, Thibault V, Cadranel JF, Bernard B, Opolon P, Coriat P, Bitker MO. Impact of hepatitis B and C virus on kidney transplantation outcome. Hepatology. 1999 Jan;29(1):257-63. doi: 10.1002/hep.510290123. PMID 9862875
- [Background] Hanafusa T, Ichikawa Y, Kishikawa H, Kyo M, Fukunishi T, Kokado Y, Okuyama A, Shinji Y, Nagano S. Retrospective study on the impact of hepatitis C virus infection on kidney transplant patients over 20 years. Transplantation. 1998 Aug 27;66(4):471-6. doi: 10.1097/00007890-199808270-00010. PMID 9734490
- [Background] Legendre C, Garrigue V, Le Bihan C, Mamzer-Bruneel MF, Chaix ML, Landais P, Kreis H, Pol S. Harmful long-term impact of hepatitis C virus infection in kidney transplant recipients. Transplantation. 1998 Mar 15;65(5):667-70. doi: 10.1097/00007890-199803150-00011. PMID 9521201
- [Background] Izopet J, Rostaing L, Sandres K, Cisterne JM, Pasquier C, Rumeau JL, Duffaut M, Durand D, Puel J. Longitudinal analysis of hepatitis C virus replication and liver fibrosis progression in renal transplant recipients. J Infect Dis. 2000 Mar;181(3):852-8. doi: 10.1086/315355. PMID 10720504
- [Background] Zylberberg H, Nalpas B, Carnot F, Skhiri H, Fontaine H, Legendre C, Kreis H, Brechot C, Pol S. Severe evolution of chronic hepatitis C in renal transplantation: a case control study. Nephrol Dial Transplant. 2002 Jan;17(1):129-33. doi: 10.1093/ndt/17.1.129. PMID 11773476
- [Background] Fabrizi F, Dulai G, Dixit V, Bunnapradist S, Martin P. Meta-analysis: interferon for the treatment of chronic hepatitis C in dialysis patients. Aliment Pharmacol Ther. 2003 Dec;18(11-12):1071-81. doi: 10.1046/j.1365-2036.2003.01780.x. PMID 14653826
- [Background] Russo MW, Goldsweig CD, Jacobson IM, Brown RS Jr. Interferon monotherapy for dialysis patients with chronic hepatitis C: an analysis of the literature on efficacy and safety. Am J Gastroenterol. 2003 Jul;98(7):1610-5. doi: 10.1111/j.1572-0241.2003.07526.x. PMID 12873587
- [Background] Kokoglu OF, Ucmak H, Hosoglu S, Cetinkaya A, Kantarceken B, Buyukbese MA, Isik IO. Efficacy and tolerability of pegylated-interferon alpha-2a in hemodialysis patients with chronic hepatitis C. J Gastroenterol Hepatol. 2006 Mar;21(3):575-80. doi: 10.1111/j.1440-1746.2005.04008.x. PMID 16638102
- [Background] Sporea I, Popescu A, Sirli R, Golea O, Totolici C, Danila M, Vernic C. Pegylated-interferon alpha 2a treatment for chronic hepatitis C in patients on chronic haemodialysis. World J Gastroenterol. 2006 Jul 14;12(26):4191-4. doi: 10.3748/wjg.v12.i26.4191. PMID 16830372
- [Background] Chan TM, Ho SK, Tang CS, Tse KC, Lam MF, Lai KN, Yung S. Pilot study of pegylated interferon-alpha 2a in dialysis patients with chronic hepatitis C virus infection. Nephrology (Carlton). 2007 Feb;12(1):11-7. doi: 10.1111/j.1440-1797.2006.00662.x. PMID 17295655
- [Background] Russo MW, Ghalib R, Sigal S, Joshi V. Randomized trial of pegylated interferon alpha-2b monotherapy in haemodialysis patients with chronic hepatitis C. Nephrol Dial Transplant. 2006 Feb;21(2):437-43. doi: 10.1093/ndt/gfi231. Epub 2005 Oct 18. PMID 16234288
- [Background] Annicchiarico BE, Siciliano M. Pegylated interferon-alpha 2b monotherapy for haemodialysis patients with chronic hepatitis C. Aliment Pharmacol Ther. 2004 Jul 1;20(1):123-4; author reply 124. doi: 10.1111/j.1365-2036.2004.01954.x. No abstract available. PMID 15225179
- [Background] Potthoff A, Wiegand J, Luth JB, Wedemeyer H, Manns MP, Tillmann HL. Superiority of standard interferon-alpha2b compared to pegylated interferon-alpha2b (12 kDa) in a hemodialysis patient with chronic hepatitis C? Clin Nephrol. 2005 Mar;63(3):232-5. doi: 10.5414/cnp63232. PMID 15786827
- [Background] Magnone M, Holley JL, Shapiro R, Scantlebury V, McCauley J, Jordan M, Vivas C, Starzl T, Johnson JP. Interferon-alpha-induced acute renal allograft rejection. Transplantation. 1995 Apr 15;59(7):1068-70. doi: 10.1097/00007890-199504150-00030. No abstract available. PMID 7709447
- [Background] Morales JM. Hepatitis C virus infection and renal disease after renal transplantation. Transplant Proc. 2004 Apr;36(3):760-2. doi: 10.1016/j.transproceed.2004.03.041. PMID 15110654
- [Background] Rostaing L, Izopet J, Baron E, Duffaut M, Puel J, Durand D. Treatment of chronic hepatitis C with recombinant alpha 2b interferon in kidney transplant recipients: preliminary results and side effects. Transplant Proc. 1995 Feb;27(1):948-50. No abstract available. PMID 7879242
- [Background] Casanovas-Taltavull T, Baliellas C, Benasco C, Serrano TT, Casanova A, Perez JL, Guerrero L, Gonzalez MT, Andres E, Gil-Vernet S, Casais LA. Efficacy of interferon for chronic hepatitis C virus-related hepatitis in kidney transplant candidates on hemodialysis: results after transplantation. Am J Gastroenterol. 2001 Apr;96(4):1170-7. doi: 10.1111/j.1572-0241.2001.03697.x. PMID 11316166
- [Background] Mousa DH, Abdalla AH, Al-Shoail G, Al-Sulaiman MH, Al-Hawas FA, Al-Khader AA. Alpha-interferon with ribavirin in the treatment of hemodialysis patients with hepatitis C. Transplant Proc. 2004 Jul-Aug;36(6):1831-4. doi: 10.1016/j.transproceed.2004.07.025. PMID 15350490
- [Background] Bruchfeld A, Stahle L, Andersson J, Schvarcz R. Ribavirin treatment in dialysis patients with chronic hepatitis C virus infection--a pilot study. J Viral Hepat. 2001 Jul;8(4):287-92. doi: 10.1046/j.1365-2893.2001.00300.x. PMID 11454181
- [Background] Bruchfeld A, Stahle L, Andersson J, Schvarcz R. Interferon and ribavirin therapy in dialysis patients with chronic hepatitis C. Nephrol Dial Transplant. 2001 Aug;16(8):1729. doi: 10.1093/ndt/16.8.1729. No abstract available. PMID 11477195
- [Background] Bruchfeld A, Lindahl K, Reichard O, Carlsson T, Schvarcz R. Pegylated interferon and ribavirin treatment for hepatitis C in haemodialysis patients. J Viral Hepat. 2006 May;13(5):316-21. doi: 10.1111/j.1365-2893.2005.00680.x. PMID 16637862
- [Background] Shiffman ML, Di Bisceglie AM, Lindsay KL, Morishima C, Wright EC, Everson GT, Lok AS, Morgan TR, Bonkovsky HL, Lee WM, Dienstag JL, Ghany MG, Goodman ZD, Everhart JE; Hepatitis C Antiviral Long-Term Treatment Against Cirrhosis Trial Group. Peginterferon alfa-2a and ribavirin in patients with chronic hepatitis C who have failed prior treatment. Gastroenterology. 2004 Apr;126(4):1015-23; discussion 947. doi: 10.1053/j.gastro.2004.01.014. PMID 15057741

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: June 2006- June 2007 Location: 5 academic centers
Pre-assignment Details: Wash out period: 6 months after last interferon intervention
Groups:
- Pegylated Interferon and Ribavirin for 48 Weeks (Genotype 1): Pegylated interferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 135 ug/week plus ribavirin (Copegus, F. Hoffman-LaRoche) 200 mg/day for 48 weeks
- Pegylated Interferon and Ribavirin for 24 Weeks (Genotype 2): Pegylated interferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 135 ug/week plus ribavirin (Copegus, F. Hoffman-LaRoche) 200 mg/day for 24 weeks
Period: Overall Study
Arm/Group | Pegylated Interferon and Ribavirin for 48 Weeks (Genotype 1) | Pegylated Interferon and Ribavirin for 24 Weeks (Genotype 2)
Started | 25 | 10
Completed | 18 | 8
Not Completed | 7 | 2
Not completed — Adverse Event | 5 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pegylated Interferon and Ribavirin for 48 Weeks (Genotype 1) | Pegylated Interferon and Ribavirin for 24 Weeks (Genotype 2) | Total
Number analyzed (Participants) | 25 | 10 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 10 | 35
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48 (8) | 44 (12) | 47 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 17 | 6 | 23
Region of Enrollment [Number; unit: participants]
  Taiwan | 25 | 10 | 35

OUTCOME MEASURES:

1. Primary Outcome: 1.Number of Participants With Sustained Virologic Response (SVR) 2.Number of Participants Who Droppoed Out of the Study Prematurely Due to Adverse Events (AEs)
Description: 1. Number of participants with sustained virologic response (SVR): number of patients with undetectable HCV RNA 6 months off therapy by real-time PCR test (Cobas TaqMan HCV Test v2.0, Roche Diagnostics GmbH, Mannheim, Germany, limit of detection < 25 IU/mL)
  2. Number of participants who droppoed out of the study prematurely due to adverse events (AEs): number of patients who prematurely withdrew from the study due to any adverse events
Time Frame: 1.5 year
Population: Outcome measures:intention-to-treat (ITT) analysis Imputation technique: last observation carried forward
Measure: Number; unit: Participants
Arm/Group | Pegylated Interferon and Ribavirin for 48 Weeks (Genotype 1) | Pegylated Interferon and Ribavirin for 24 Weeks (Genotype 2)
Number analyzed (Participants) | 25 | 10
Participants
  Sustained virologic response (SVR) | 13 | 8
  Drop-out | 7 | 2

2. Secondary Outcome: Number of Participants With Histologic Response(HR)
Description: Number of participants with histologic response (HR): number of patients who had improvement of as least 2 scores at the end of follow-up liver biopsy compared to baseline liver biopsy by Ishak scoring system (the sum of Ishak necroinflammation score (0-18) and Ishak fibrosis score (0-6); the higher the total scores, the severer the histologic changes)
Time Frame: 1.5 year
Measure: Number; unit: Participants
Arm/Group | Pegylated Interferon and Ribavirin for 48 Weeks (Genotype 1) | Pegylated Interferon and Ribavirin for 24 Weeks (Genotype 2)
Number analyzed (Participants) | 25 | 10
Participants | 11 | 6

ADVERSE EVENTS:
Time Frame: 18 months
Description: Constitutional symptoms and abnormal laboratory tests
Arm/Group | Pegylated Interferon and Ribavirin for 48 Weeks (Genotype 1) | Pegylated Interferon and Ribavirin for 24 Weeks (Genotype 2)
Serious Adverse Events (participants affected / at risk) | 2/25 | 1/10
Other Adverse Events (participants affected / at risk) | 22/25 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegylated Interferon and Ribavirin for 48 Weeks (Genotype 1) (N=25) | Pegylated Interferon and Ribavirin for 24 Weeks (Genotype 2) (N=10)
Optic neuritis (Eye disorders) | 1 (1) | 1 (1)
Interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegylated Interferon and Ribavirin for 48 Weeks (Genotype 1) (N=25) | Pegylated Interferon and Ribavirin for 24 Weeks (Genotype 2) (N=10)
Fever (Infections and infestations) | 6 (6) | 3 (3)
Rigor (Immune system disorders) | 6 (6) | 2 (2)
Fatigue (Nervous system disorders) | 14 (14) | 8 (8)
Headache (Nervous system disorders) | 7 (7) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Arthralgia (Immune system disorders) | 1 (1) | 1 (1)
Insomnia (Nervous system disorders) | 7 (7) | 4 (4)
Irritability (Nervous system disorders) | 2 (2) | 1 (1)
Depression (Nervous system disorders) | 3 (3) | 1 (1)
Anorexia (Gastrointestinal disorders) | 5 (5) | 5 (5)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Body weight loss (General disorders) | 3 (3) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Aphthous ulcer (Immune system disorders) | 4 (4) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nasal stuffiness (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 20 (20) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No